CLINICAL TRIAL: NCT03867981
Title: Phone Coaching and Internet-delivered Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1296020; 5R01DK117843 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-08 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: Obesity; weight loss; exercise; diet; phone coaching
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet weight loss + possibility of brief phone coaching (Experimental): Participants randomized to this group will receive a 4-month, Internet-delivered weight loss program followed by an 8-month, Internet-delivered weight loss maintenance program. All individuals will be taught behavioral strategies for changing diet and physical activity behaviors via video lessons. Some participants in this group will also be selected to receive a brief period (i.e., once/week for 3 weeks) of phone coaching starting at week 5. The first coaching call will be approximately 45 minutes in duration and remaining calls with be 10-15 minutes. Coaches will problem solve with participants and help them develop an individualized meal plan.
  Interventions: Behavioral: Internet-based weight loss program; Behavioral: Brief phone coaching
- Internet weight loss + possibility of extended phone coaching (Experimental): Participants randomized to this group will receive a 4-month, Internet-delivered weight loss program followed by an 8-month, Internet-delivered weight loss maintenance program. All individuals will be taught behavioral strategies for changing diet and physical activity behaviors via video lessons. Some participants in this group will also be selected to receive an extended period (i.e., once/week for 12 weeks) of phone coaching starting at week 5. The first coaching call will be approximately 45 minutes in duration and remaining calls with be 10-15 minutes. Coaches will problem solve with participants and help them develop an individualized meal plan.
  Interventions: Behavioral: Internet-based weight loss program; Behavioral: Extended phone coaching
- Internet weight loss only (Active Comparator): Participants randomized to this group will receive a 4-month, Internet-delivered weight loss program followed by an 8-month, Internet-delivered weight loss maintenance program. All individuals will be taught behavioral strategies for changing diet and physical activity behaviors via video lessons. No participants in this group will receive any phone coaching.
  Interventions: Behavioral: Internet-based weight loss program

INTERVENTIONS:
Behavioral: Internet-based weight loss program — 12-month, Internet-based weight loss/maintenance program.
Behavioral: Brief phone coaching — Some individuals will receive 3 weeks of phone coaching. Coaching calls will occur 1x/week, starting at week 5. Once coaching calls are completed, the participant will not have any other contact with their coach.
  Arms: Internet weight loss + possibility of brief phone coaching
Behavioral: Extended phone coaching — Some individuals will receive 12 weeks of phone coaching. Coaching calls will occur 1x/week, starting at week 5. Once coaching calls are completed, the participant will not have any other contact with their coach.
  Arms: Internet weight loss + possibility of extended phone coaching

SUMMARY:
The purpose of this study is to examine whether adding phone coaching to an Internet-based weight loss program can improve weight loss outcomes at 4 months and 1 year. All individuals will receive a 4-month, Internet-delivered weight loss program followed by an 8-month Internet-delivered weight loss maintenance program. Some individuals will also be selected to receive either 3 weeks or 12 weeks of phone coaching. Assessments of weight, diet, physical activity, and psychosocial factors will occur at baseline, 4 months, and 1 year.

DETAILED DESCRIPTION:
All individuals enrolled in this study will receive a 4-month Internet-based weight loss program followed by an 8-month Internet-based weight loss maintenance program. During the first 4 months, each week individuals will be asked to view a 10-15-minute multi-media lesson (one per week). These lessons focus on behavioral principles for changing diet and physical activity behaviors. Participants are also given weight loss, calorie intake, and physical activity goals. They are taught how to self-monitor this information and are instructed to submit it weekly on the study website. Automated, weekly individualized feedback is provided. Following the 4-month weight loss program participants will receive an 8-month weight loss maintenance program. During this time, they will be asked to view monthly video lessons which focus on strategies for successful WL maintenance and instructed to continue to self-monitor weight, calorie intake, and physical activity minutes on the study website for one week per month. Automated, monthly feedback is provided.

In addition to the Internet program described above, some individuals enrolled in this study will be selected to receive phone coaching. Those selected for 'brief' phone coaching will be asked to complete 3 phone calls with a coach between weeks 5-8 of the study and those selected to receive 'extended' phone coaching will be asked to complete 12 phone calls with a coach between weeks 5-16. The first coaching call will be approximately 45 minutes in duration and all subsequent calls will be approximately 15 minutes in duration. The coach will assist participants in developing a meal plan, problem solving around current barriers, and goal setting. Upon completion of all coaching calls participants will have no additional interaction with the coach, but will remain enrolled in the Internet program.

Assessments will occur at baseline, 4, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* BMI: 25-45 kg/m2
* Regular internet access

Exclusion Criteria:

* Currently pregnant, <6 months post-partum, nursing, or planning to become pregnant within the next 12 months.
* Current enrollment in a commercial weight loss program or other weight loss research study
* Currently taking weight loss medications
* Previously had bariatric surgery
* Inability to walk 2 blocks without stopping
* Any medical condition for which weight loss, dietary restriction, or physical activity is contraindicated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Unick, PhD, Principal Investigator — The Miriam Hospital's Weight Control and Diabetes Research Center
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, and informed consent document can be found within this clinicaltrials.gov record. Requests to view or utilize de-identified, participant-level data can be sent to the Principal Investigator (Dr. Jessica Unick - junick@lifespan.org).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: baseline to 12 months
Access Criteria: Requests to view or utilize de-identified, participant-level data can be sent to the Principal Investigator (Dr. Jessica Unick - junick@lifespan.org).

REFERENCES:
- [Derived] Unick JL, Pellegrini CA, Dunsiger SI, Demos KE, Thomas JG, Bond DS, Lee RH, Webster J, Wing RR. An Adaptive Telephone Coaching Intervention for Patients in an Online Weight Loss Program: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2414587. doi: 10.1001/jamanetworkopen.2024.14587. PMID 38848067

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization occurred at baseline, but participants were not informed of their randomization assignment until 1 month. Those reporting a 1-month weight then went on to receive brief coaching, extended coaching, or no coaching based upon randomization assignment.
Period: Overall Study
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Started | 150 | 150 | 152
Reported Weight at 1 Month | 143 | 148 | 146
Completed 4-month Assessment | 134 | 135 | 126
Completed | 131 | 131 | 115
Not Completed | 19 | 19 | 37

BASELINE CHARACTERISTICS:
Population: These data only include participants who reported a 1-month weight (n=437 out of 452 who began the weight loss program), given that those who did not report a 1-month weight were not eligible to receive coaching and did not continue with the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only | Total
Number analyzed (Participants) | 143 | 148 | 146 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.5) | 50.7 (10.9) | 48.5 (11.4) | 50.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 101 | 103 | 305
  Male | 42 | 47 | 43 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 23 | 56
  Not Hispanic or Latino | 128 | 130 | 123 | 381
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants who selected 'other' for race were coded as 'unknown or not reported'
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 2 | 3 | 2 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 15 | 10 | 14 | 39
    White | 115 | 119 | 114 | 348
    More than one race | 4 | 5 | 3 | 12
    Unknown or Not Reported | 7 | 11 | 13 | 31
Region of Enrollment [Number; unit: participants]
  United States | 143 | 148 | 146 | 437

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change at 4 Months
Description: Weight change was assessed using weight at baseline and 4 months
Time Frame: 4 months after start of weight loss program
Population: Reflects the number of participants in each treatment arm who completed the 4-month assessment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Number analyzed (Participants) | 134 | 135 | 126
percent change | -6.2 (4.7) | -7.0 (5.1) | -4.5 (4.7)

2. Primary Outcome: Percent Weight Change at 12 Months
Description: Weight change was assessed using weight at baseline and 12 months
Time Frame: 12 months after start of weight loss program
Population: Reflects the number of participants who completed the 12-month assessment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Number analyzed (Participants) | 131 | 131 | 115
percent change | -4.9 (6.1) | -5.5 (6.7) | -3.9 (7.4)

3. Secondary Outcome: Cost of Supplemental Coaching Per kg of Weight Loss
Description: Cost-effectiveness analyses were completed to determine the intervention cost per kg of weight loss
Time Frame: 12 months after start of weight loss program
Population: The cost of adding supplemental coaching to a pre-existing weight loss program was calculated per enrolled participant. Data was not collected in the "Internet Weight Loss Only" Arm for this outcome measure since these participants did not receive supplemental coaching.
Measure: Number; unit: dollars per kilogram of weight loss
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching
Number analyzed (Participants) | 150 | 150
dollars per kilogram of weight loss | 13.2 | 30.8

4. Secondary Outcome: Change in Physical Activity Minutes (Min/wk)
Description: Physical activity was assessed via Actigraph accelerometers and included moderate-to-vigorous physical activity that was accumulated in bouts of >=10 minutes. A change score between baseline and 4 months was calculated.
Time Frame: 4 months after study enrollment
Population: The participant flow data for this study was based upon whether or not weight (the primary outcome) was measured at each assessment period. Some participants completed a weight assessment at 4 months but either did not wear the physical activity monitor or did not wear the monitor for enough days (i.e., 4 or more days with greater than 8 hours of device wear time per day). Thus, the number of participants analyzed here is less than what was reported in the Participant Flow.
Measure: Mean (Standard Deviation); unit: change in min/wk
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Number analyzed (Participants) | 123 | 124 | 109
change in min/wk | 55.37 (106.82) | 44.45 (108.43) | 24.01 (94.43)

5. Secondary Outcome: Change in Dietary Intake (Kcals)
Description: Dietary intake was assessed using self-reported kcal totals obtained from food diaries. The change was calculated from baseline to 4 months.
Time Frame: 4 months after start of weight loss program
Population: The participant flow data for this study was based upon whether or not weight (the primary outcome) was measured at each assessment period. Some participants completed a weight assessment at 4 months but did not complete a food diary at this time point. Thus, the number of participants analyzed here is less than what was reported in the Participant Flow.
Measure: Mean (Standard Deviation); unit: change in kcals
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Number analyzed (Participants) | 111 | 111 | 97
change in kcals | -417.78 (379.62) | -528.51 (389.79) | -500.51 (401.76)

6. Secondary Outcome: Self-monitoring of Calorie Intake
Description: Percentage of days that participant self-monitored their calorie intake on study website
Time Frame: 4 months after start of weight loss program
Population: Percentage of days that participants monitored their calorie intake on the study website over the first 4 months of the program (out of 112)
Measure: Mean (Standard Deviation); unit: % of days
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Number analyzed (Participants) | 134 | 135 | 126
% of days | 79.5 (27.3) | 85.4 (23.4) | 66.5 (31.4)

7. Secondary Outcome: Video Lesson Viewing
Description: Percentage of video lessons viewed on study website
Time Frame: 4 months after start of weight loss program
Population: Percentage of weekly video lessons that participants viewed over the first 4 months of the program (out of 16)
Measure: Mean (Standard Deviation); unit: % of lessons
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
Number analyzed (Participants) | 134 | 135 | 126
% of lessons | 68.7 (28.9) | 83.0 (26.6) | 52.0 (32.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entire 12-month intervention period
Arm/Group | Internet Weight Loss + Possibility of Brief Phone Coaching | Internet Weight Loss + Possibility of Extended Phone Coaching | Internet Weight Loss Only
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/148 | 0/146
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/148 | 0/146
Other Adverse Events (participants affected / at risk) | 0/143 | 0/148 | 0/146

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT03867981/Prot_SAP_001.pdf
  • Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03867981/ICF_000.pdf